CLINICAL TRIAL: NCT01743118
Title: Phase Ib, Two-centre, Randomised, Observer-blind, Placebo- and Comparator Controlled Trial to Evaluate the Safety, Tolerability and Antipsoriatic Efficacy of Three Strengths of a Topical SPS4251 Formulation in a Psoriasis Plaque Test
Brief Title: Antipsoriatic Effect of a Topical Formulation for the Treatment of Psoriasis Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Bioskin GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SP001
Record Dates: First submitted 2012-12-03; First posted 2012-12-06 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psoriasis Plaque Test (Experimental): SPS4251 Ointment, 0.01%; SPS4251 Ointment, 0.1%; SPS4251 Ointment, 1%; SPS4251 Placebo, Daivonex® ointment
  Interventions: Drug: SPS4251 Ointment; Drug: Placebo; Drug: Daivonex® ointment

INTERVENTIONS:
Drug: SPS4251 Ointment — Approximately 200 µl of each TREATMENT will be topically applied per test field (1.1 cm2) once daily during a 12-day treatment period (10 treatments)
Drug: Placebo — Approximately 200 µl of each TREATMENT will be topically applied per test field (1.1 cm2) once daily during a 12-day treatment period (10 treatments)
Drug: Daivonex® ointment — Approximately 200 µl of each TREATMENT will be topically applied per test field (1.1 cm2) once daily during a 12-day treatment period (10 treatments).
  Other Names: calcipotriol

SUMMARY:
The current most important topical treatments for psoriasis are vitamin D3 analogues and/or corticosteroids. The possibility of another effective treatment for psoriasis could be based on the immunosuppressive efficacy of selective blockers of a lymphocyte potassium channel.

The aim of the clinical trial is to evaluate the safety, tolerability and anti-psoriatic efficacy of topical SPS4251 formulations in comparison to placebo and to a marketed topical Vitamin-D analogue ointment in a psoriasis plaque test.

ELIGIBILITY:
Inclusion Criteria:

* men aged 18 years or older
* subjects with mild to moderate psoriasis vulgaris in a chronic stable phase
* subject with up to three stable plaques with an area sufficient for five treatment fields
* Plaques to be treated should have a comparable thickness of the Echo Lucent Band of at least 200 µm

Exclusion Criteria:

* Subjects with guttate psoriasis, punctate psoriasis, erythrodermic psoriasis, psoriatic arthropathy and pustular psoriasis
* Local treatment with antipsoriatics in the 4 weeks preceding and/or during the trial, and any topical antipsoriatic treatment on the plaques to be treated in this trial in the 8 weeks before first treatment and/or during the trial
* Systemic treatment with antipsoriatics e.g. corticosteroids, cytostatics, retinoids in the three months before first treatment and during the trial;
* Treatment with systemic medications or medications acting locally which might have countered or influenced the trial aim
* Contraindications according to summary of product characteristics of Daivonex® Ointment;
* UV-therapy within four weeks before first treatment and during the trial
* Symptoms of a clinically significant illness that may influence the outcome of the trial in the four weeks before baseline visit and during the trial
* Any history of cardiovascular disease
* Any evidence of ECG abnormality on screening ECG
* Close affiliation with the Investigator (e.g. a close relative) or persons working at bioskin GmbH or subject is an employee of the Sponsor;
* Subject is institutionalized because of legal or regulatory order.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of plaque thickness-reducing efficacy measured by 20 MHz sonography of psoriatic infiltrate | Up to Day 12

SECONDARY OUTCOMES:
Evaluation of anti-psoriatic efficacy by clinical assessment | Up to day 12
Number of subjects with Adverse Events | Up to day 12

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Bioskin, Berlin
  - Bioskin, Hamburg